CLINICAL TRIAL: NCT05805813
Title: Cross-control Study on the Effect of Peritoneal Rest on Peritoneal Transport Function in Peritoneal Dialysis Patients
Acronym: CSEPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Wu Bei, Principal Investigator, Peking University People's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: peritoneal rest trial
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Disease 5D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): group A carry on continuous ambulatory peritoneal dialysis (the original dialysis method) for 1 month, and then changed to intermittent peritoneal dialysis at night (using automatic peritoneal dialysis machine) for 1 month
  Interventions: Combination Product: peritoneal rest
- Group B (Experimental): Group B carry on intermittent peritoneal dialysis at night (using automatic peritoneal dialysis machine) for 1 month, and then change to continuous ambulatory peritoneal dialysis (original dialysis method) for 1 month.
  Interventions: Combination Product: peritoneal rest

INTERVENTIONS:
Combination Product: peritoneal rest — Change continuous ambulatory peritoneal dialysis to intermittent peritoneal dialysis at night (using automatic peritoneal dialysis machine) for 1 month. In this way, give a chance of peritoneum rest.

SUMMARY:
The investigators will carry out a prospective cross-over, pre-and post-controlled clinical study : 36 patients with continuous ambulatory peritoneal dialysis with high/high average transport will be recruited and treated with continuous ambulatory peritoneal dialysis and intermittent peritoneal dialysis at night (using automatic peritoneal dialysis machine) for 1 month respectively. The changes of peritoneal transport function and ultrafiltration volume before and after the two dialysis methods will be compared.

DETAILED DESCRIPTION:
1. Inclusion Criteria

   * Continuous ambulatory peritoneal dialysis for more than 3 months;
   * The peritoneal transport function is high/high average transport (D/Pcr>0.65 at 4 hours in the peritoneal balance test);
   * Sign the informed consent form voluntarily.
2. Exclusion Criteria

   * Patients with peritonitis in the past 3 months;
   * Patients with acute complications such as cardiovascular events, pulmonary infection and gastrointestinal bleeding in the past 3 months;
   * The doctor judged that it was not suitable for the patients in this study for other reasons.
3. Treatment plan

   The patients will be divided into two groups randomly: group A carry on continuous ambulatory peritoneal dialysis (the original dialysis plan) for 1 month, and then changed to intermittent peritoneal dialysis at night (using automatic peritoneal dialysis machine，the concentration and dosage of dialysate are consistent with the original plan) for 1 month; Group B carry on intermittent peritoneal dialysis at night (using automatic peritoneal dialysis machine，the concentration and dosage of dialysate are consistent with the original plan) for 1 month, and then change to continuous ambulatory peritoneal dialysis (original dialysis plan) for 1 month.
4. Observation indicators

Main observation indicators:

Changes in peritoneal transport rate (represented by 4-hour D/Pcr in the standard peritoneal balance test) and ultrafiltration volume (represented by 4-hour ultrafiltration volume in the standard peritoneal balance test) before and after daytime dry abdomen (intermittent peritoneal rest) and continuous peritoneal dialysis.

Secondary outcome measures:

changes in IL-1, IL-6 and TNF- α， VEGF and CTGF of the exudate in the standard peritoneal balance test before and after daytime dry abdomen (intermittent peritoneal rest) and continuous peritoneal dialysis .

Changes of body weight, blood pressure, hemoglobin, albumin, calcium, phosphorus, electrolyte, urea clearance index, etc. before and after daytime dry abdomen (intermittent peritoneal rest) and continuous peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria：

* Continuous ambulatory peritoneal dialysis for more than 3 months;
* The peritoneal transport function is high/high average transport (D/Pcr>0.65 at 4 hours in the peritoneal balance test);
* Sign the informed consent form voluntarily.

Exclusion criteria：

* Patients with peritonitis in the past 3 months;
* Patients with acute complications such as cardiovascular events, pulmonary infection and gastrointestinal bleeding in the past 3 months;
* The doctor judged that it was not suitable for the patients in this study for other reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
peritoneal transport rate | 1 month
  represented by 4-hour D/Pcr in the standard peritoneal balance test
ultrafiltration volume | 1 month
  represented by 4-hour ultrafiltration volume in the standard peritoneal balance test

CONTACTS AND LOCATIONS:
Overall Officials: Li Zuo, Doctor, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Twardowski ZJ. Clinical value of standardized equilibration tests in CAPD patients. Blood Purif. 1989;7(2-3):95-108. doi: 10.1159/000169582. PMID 2663040
- [Result] Maksic D, Vasilijic S, Colic M, Stankovic-Popovic V, Bokonjic D. Systemic and intraperitoneal proinflammatory cytokine profiles in patients on continuous ambulatory peritoneal dialysis. Adv Perit Dial. 2009;25:50-5. PMID 19886317
- [Result] Toda N, Mori K, Kasahara M, Koga K, Ishii A, Mori KP, Osaki K, Mukoyama M, Yanagita M, Yokoi H. Deletion of connective tissue growth factor ameliorates peritoneal fibrosis by inhibiting angiogenesis and inflammation. Nephrol Dial Transplant. 2018 Jun 1;33(6):943-953. doi: 10.1093/ndt/gfx317. PMID 29165602